CLINICAL TRIAL: NCT04311957
Title: A Randomized Non-Inferiority Trial to Compare the Efficacy of Switching From Protease-Inhibitor Based Second-Line Therapy to Bictegravir-Tenofovir Alafenamide-Emtricitabine in Virologically Suppressed Adults in Haiti
Brief Title: Continuation of Protease-Inhibitor Based Second-Line Therapy vs. Switch to B/F/TAF in Virologically Suppressed Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other)
Collaborators: Brigham and Women's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); Analysis Group, Inc. (Industry); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-US-380-5733
Record Dates: First submitted 2020-03-15; First posted 2020-03-17 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: HIV-1-infection; Antiretroviral Therapy
Keywords: HIV; Second-line therapy; Integrase strand transfer inhibitor; Protease inhibitor

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the B/F/TAF or continuation bPI group in a 1:1 ratio.
Masking Description: Open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Boosted PI Group (Active Comparator): Continuation of the same second-line regimen taken prior to entry:
  This includes either Lopinavir/ritonavir (LPVr) 400 mg/100 mg BID or Atazanavir/ritonavir (ATV/r) 300 mg/100 mg QD
  plus 2 nucleoside reverse transcriptase inhibitors (NRTIs).
  Interventions: Drug: Continuation of boosted PI
- B/F/TAF Group (Experimental): Combination tablet of bictegravir 50 mg/emtricitabine 200 mg/tenofovir alafenamide 25 mg (B/F/TAF) administered orally, once daily.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: Continuation of boosted PI — Continuation of the same second-line regimen taken prior to entry:
  LPVr 400 mg/100 mg BID or ATVr 300 mg/100 mg QD + 2 NRTIs
  Arms: Boosted PI Group
Drug: B/F/TAF — Single-tablet, fixed dose combination of bictegravir 50 mg/emtricitabine 200 mg/tenofovir alafenamide 25 mg (B/F/TAF) administered orally, once daily.
  Arms: B/F/TAF Group

SUMMARY:
This randomized trial compares the efficacy of switching to a fixed-dose combination of B/F/TAF versus continuing a boosted protease inhibitor (bPI) regimen in HIV-1 infected participants who are virologically suppressed (HIV-1 RNA <200 copies) on a second-line bPI regimen. Half of participants will receive B/F/TAF and half will continue a bPI regimen. The hypothesize is that B/F/TAF will have efficacy that is non-inferior to the boosted PI regimen.

DETAILED DESCRIPTION:
The second generation integrase strand transfer inhibitors (INSTIs) dolutegravir (DTG) and bictegravir (BIC) are widely prescribed for the treatment of HIV, due to their favorable tolerability and toxicity profile, durable efficacy, and high barrier to resistance. However, there are limited data to guide the management of patients who are already virally suppressed on a second-line bPI regimen.

Though bPIs have a high barrier to resistance and durable virologic efficacy, they have several important drug-drug interactions, are associated with unfavorable long-term metabolic effects, and may be poorly tolerated. For these reasons, a second-generation INSTI would be preferable to a boosted PI regimen, as long INSTIs are demonstrated to have non-inferior efficacy for patients who are already suppressed on a second-line bPI regimen.

In the proposed study, the efficacy of continuing the bPI regimen will be compared to switching to B/F/TAF.

ELIGIBILITY:
Inclusion Criteria:

* The ability and willingness to give informed consent.
* Age ≥18 years
* History of meeting WHO criteria for immunologic or virologic failure after receipt of a first-line treatment regimen for ≥6 months
* Currently receiving a second-line ART regimen including either ATVr or LPVr + 2 NRTIs for ≥6 months
* At least one HIV-1 RNA <200 copies/mL within 12 months prior to enrollment, and no HIV-1 RNA of at least 200 copies/mL during this period.
* Plasma HIV-1 RNA <200 copies/mL at Screening Visit.
* eGFR ≥ 50 mL/min according to the MDRD study equation for creatinine clearance
* Hepatic transaminases (AST and ALT) </=5X upper limit of normal (ULN)
* No active TB
* Women of childbearing age must agree to take reliable contraception

Exclusion Criteria:

* Active World Health Organization Stage 3 or 4 condition
* Treatment with an INSTI in the past
* Gap in care of at least one month in the prior six months
* Current alcohol or substance use judged by investigator to potentially interfere with participant study compliance
* History of poor adherence, that in the opinion of the investigator, would potentially interfere with study compliance
* Pregnant or breastfeeding at screening visit
* Planning to transfer care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Virologic failure - 200 Copies/mL cut-off | Week 48
  Proportion of participants with HIV-1 RNA at least 200 copies/mL at Week 48 as defined by the US FDA-defined snapshot algorithm

SECONDARY OUTCOMES:
Virologic failure - 50 Copies/mL cut-off | Week 48
  Proportion of participants with HIV-1 RNA at least 50 copies/mL at Week 48 as defined by the US FDA-defined snapshot algorithm
Virologic failure - 1000 Copies/mL cut-off | Week 48
  Proportion of participants with HIV-1 RNA at least 1000 copies/mL at Week 48 as defined by the US FDA-defined snapshot algorithm
Tolerability as measured by discontinuing medication | Entry to 48 weeks
  Proportion of participants discontinuing therapy for drug-related adverse events
Adverse events | Entry to 48 weeks
  Proportion of participants with 1 or more NIH Division of AIDS Grade 3 or 4 adverse events (at least 1 grade increase from baseline)
Change in cholesterol | Entry to 48 weeks
  Median change in cholesterol
Change in weight | Entry to 48 weeks
  Median change in weight in kilograms
Change in body mass index | Entry to 48 weeks
  Median change in body mass index (weight in kilograms divided by the square of height in meters)
Weight gain of 10% or greater | Entry to 48 weeks
  Proportion of participants with weight gain of at least 10% (in kilograms)
Change in waist circumference | Entry to 48 weeks
  Median change in waist circumference
Waist to hip ratio | Entry to 48 weeks
  Median change in waist to hip ratio
Adherence | Entry to 48 weeks
  Median adherence as measured by pharmacy refill records

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Severe, MD, Principal Investigator — Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic; Serena Koenig, MD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- GHESKIO, Port-au-Prince, Haiti

REFERENCES:
- [Derived] Severe P, Pierre S, Homeus F, Marc JB, Trevisi L, Aristhomene ML, Bernadin GR, Lavoile K, Rivera V, Duchatellier CF, Joseph MJ, Wu J, Rouzier V, Preval F, Jean E, Bernadin J, Zion A, Pierre Louis Forestal G, Avila-Rios S, Garcia Morales C, Zhang A, Israelski D, Apollon A, Dumont E, Fox E, Cremieux PY, Pape JW, Collins SE, Liautaud B, Sax PE, Koenig SP. Bictegravir, emtricitabine, and tenofovir alafenamide versus ritonavir-boosted protease inhibitor-based antiretroviral therapy in people with HIV and viral suppression on second-line therapy in Haiti: an open-label, randomised, non-inferiority trial. Lancet HIV. 2025 Sep;12(9):e616-e626. doi: 10.1016/S2352-3018(25)00130-4. PMID 40883049